CLINICAL TRIAL: NCT03728569
Title: Skin Barrier Dysfunction and the Role of Skin Barrier Restoration on Cutaneous and Systemic Inflammation in the Aged Population
Brief Title: Skin Barrier Dysfunction and the Role of Skin Barrier Restoration
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment and interactions/interventions paused due to COVID-19. Not expected to resume in the future. This is not a suspension of IRB approval
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Gary Fisher, Professor, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00138533 / Derm 719
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Cutaneous Inflammation
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Intervention Model Description: Both groups, young and old, will receive the same intervention; therefore, single group study model was chosen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects over the age of 70 yrs receiving Vanicream (Other): Subjects will be instructed to apply a moisturizer over the entire skin surface from the neck down twice daily. Subjects will also be required to use a bar soap (Vanicream Cleansing Bar) once daily and avoid application of other soaps or cleaners to the body for the duration of the study.
  Interventions: Other: Vanicream Moisturizing Skin Cream; Other: Vanicream Cleansing Soap
- Subjects between 18 and 30 yrs receiving Vanicream (Other): Subjects will be instructed to apply a moisturizer over the entire skin surface from the neck down twice daily. Subjects will also be required to use a bar soap (Vanicream Cleansing Bar) once daily and avoid application of other soaps or cleaners to the body for the duration of the study.
  Interventions: Other: Vanicream Moisturizing Skin Cream; Other: Vanicream Cleansing Soap

INTERVENTIONS:
Other: Vanicream Moisturizing Skin Cream — Vanicream Moisturizing Skin Cream daily application
Other: Vanicream Cleansing Soap — Vanicream Cleansing Soap daily use

SUMMARY:
The objective of this exploratory study is to gain an understanding of cutaneous and systemic inflammation and how restoration of the skin barrier through the use of moisturizer may restore the skin barrier function and reduce systemic inflammation in elderly humans compared to the young. The exploratory study will consist of three visits per subject. Subjects will be instructed to apply a moisturizer (Vanicream Moisturizing Skin Cream) over the entire skin surface from the neck down twice daily for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

Aged group (>70 years old)

* In good general health
* Body mass index (BMI) preferably in the healthy range (approximately 25 kg/m2) and no greater than 30 kg/m2
* Fitzpatrick skin types I-V
* Disrupted skin barrier defined as transepidermal water loss (TEWL) >5 g/m2/h on the upper arms or >3 g/m2/h on the buttocks
* Clinical signs of skin dryness as determined by the investigator.
* No disease states or physical conditions that would impair evaluation of the biopsy sites
* Signed, written and witnessed informed consent form
* Willing to comply with study procedures

Young group (18-30 years old)

* Good general health
* BMI preferably in the healthy range (approximately 25 kg/m2) and no greater than 30 kg/m2
* Fitzpatrick skin types I-V
* Disrupted skin barrier defined as transepidermal water loss (TEWL) >5 g/m2/h on the upper arms or >3 g/m2/h on the buttocks
* Clinical signs of skin dryness as determined by the investigator
* No disease states or physical conditions that would impair evaluation of the biopsy sites
* Signed, written and witnessed informed consent form
* Willing to comply with study procedures

Exclusion Criteria:

* Pregnant or lactating women or women contemplating pregnancy for the duration of the protocol (determined by self-report; if subjects are unsure of their pregnancy status, they will be excluded).
* Frailty as determined by research study nurse
* History of inflammatory skin conditions such as psoriasis or atopic dermatitis.
* History of uncontrolled inflammatory or autoimmune disease.
* History of keloids or any other condition that would complicate wound healing
* History of allergic reactions to local lidocaine
* Frequent nonsteroidal anti-inflammatory drug (NSAID) use (not including low dose aspirin) and unwilling/unable to discontinue NSAIDS for 2 weeks prior to enrollment to the end of the study.
* Systemic steroids (excluding inhaled steroids for asthma) and unwilling/unable to discontinue systemic steroids for 3 weeks prior to enrollment to the end of the study.
* Topical corticosteroid use within 2 weeks of enrollment.
* Topical immunomodulation use such as calcineurin inhibitors within 2 weeks of enrollment
* Other anti-inflammatory or immunodulatory medications (immunosuppression)
* Received an experimental drug or used an experimental device 30 days prior to admission to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in skin hydration status in aged and young subjects | up to 30 days
  Trans-epidermal water loss (TEWL) will be performed on the upper arm and buttocks at Visits 1 and 2. This instrument will measure the amount of water that is lost through the skin. The change in skin hydration status in each subject will be assessed and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Fisher, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghadially R, Brown BE, Sequeira-Martin SM, Feingold KR, Elias PM. The aged epidermal permeability barrier. Structural, functional, and lipid biochemical abnormalities in humans and a senescent murine model. J Clin Invest. 1995 May;95(5):2281-90. doi: 10.1172/JCI117919. PMID 7738193
- [Background] White-Chu EF, Reddy M. Dry skin in the elderly: complexities of a common problem. Clin Dermatol. 2011 Jan-Feb;29(1):37-42. doi: 10.1016/j.clindermatol.2010.07.005. PMID 21146730
- [Background] Kim HO, Kim HS, Youn JC, Shin EC, Park S. Serum cytokine profiles in healthy young and elderly population assessed using multiplexed bead-based immunoassays. J Transl Med. 2011 Jul 20;9:113. doi: 10.1186/1479-5876-9-113. PMID 21774806
- [Background] Mariani E, Cattini L, Neri S, Malavolta M, Mocchegiani E, Ravaglia G, Facchini A. Simultaneous evaluation of circulating chemokine and cytokine profiles in elderly subjects by multiplex technology: relationship with zinc status. Biogerontology. 2006 Oct-Dec;7(5-6):449-59. doi: 10.1007/s10522-006-9060-8. PMID 16967203
- [Background] Surmi BK, Hasty AH. Macrophage infiltration into adipose tissue: initiation, propagation and remodeling. Future Lipidol. 2008;3(5):545-556. doi: 10.2217/17460875.3.5.545. PMID 18978945
- [Background] Katoh N, Hirano S, Kishimoto S, Yasuno H. Acute cutaneous barrier perturbation induces maturation of Langerhans' cells in hairless mice. Acta Derm Venereol. 1997 Sep;77(5):365-9. doi: 10.2340/0001555577365369. PMID 9298129
- [Background] Lin TK, Man MQ, Santiago JL, Park K, Roelandt T, Oda Y, Hupe M, Crumrine D, Lee HJ, Gschwandtner M, Thyssen JP, Trullas C, Tschachler E, Feingold KR, Elias PM. Topical antihistamines display potent anti-inflammatory activity linked in part to enhanced permeability barrier function. J Invest Dermatol. 2013 Feb;133(2):469-78. doi: 10.1038/jid.2012.335. Epub 2012 Sep 27. PMID 23014339
- [Background] Nishijima T, Tokura Y, Imokawa G, Seo N, Furukawa F, Takigawa M. Altered permeability and disordered cutaneous immunoregulatory function in mice with acute barrier disruption. J Invest Dermatol. 1997 Aug;109(2):175-82. doi: 10.1111/1523-1747.ep12319282. PMID 9242504
- [Background] Onoue A, Kabashima K, Kobayashi M, Mori T, Tokura Y. Induction of eosinophil- and Th2-attracting epidermal chemokines and cutaneous late-phase reaction in tape-stripped skin. Exp Dermatol. 2009 Dec;18(12):1036-43. doi: 10.1111/j.1600-0625.2009.00899.x. PMID 19558500
- [Background] Proksch E, Brasch J, Sterry W. Integrity of the permeability barrier regulates epidermal Langerhans cell density. Br J Dermatol. 1996 Apr;134(4):630-8. PMID 8733362
- [Background] Tsai JC, Feingold KR, Crumrine D, Wood LC, Grunfeld C, Elias PM. Permeability barrier disruption alters the localization and expression of TNF alpha/protein in the epidermis. Arch Dermatol Res. 1994;286(5):242-8. doi: 10.1007/BF00387595. PMID 8060154
- [Background] Wood LC, Stalder AK, Liou A, Campbell IL, Grunfeld C, Elias PM, Feingold KR. Barrier disruption increases gene expression of cytokines and the 55 kD TNF receptor in murine skin. Exp Dermatol. 1997 Apr;6(2):98-104. doi: 10.1111/j.1600-0625.1997.tb00154.x. PMID 9209892
- [Background] Hu L, Mauro TM, Dang E, Man G, Zhang J, Lee D, Wang G, Feingold KR, Elias PM, Man MQ. Epidermal Dysfunction Leads to an Age-Associated Increase in Levels of Serum Inflammatory Cytokines. J Invest Dermatol. 2017 Jun;137(6):1277-1285. doi: 10.1016/j.jid.2017.01.007. Epub 2017 Jan 20. PMID 28115059
- [Background] Jiang YJ, Lu B, Crumrine D, Man MQ, Elias PM, Feingold KR. IL-1alpha accelerates stratum corneum formation and improves permeability barrier homeostasis during murine fetal development. J Dermatol Sci. 2009 May;54(2):88-98. doi: 10.1016/j.jdermsci.2009.01.001. Epub 2009 Feb 11. PMID 19216058
- [Background] Jung YJ, Jung M, Kim M, Hong SP, Choi EH. IL-1alpha stimulation restores epidermal permeability and antimicrobial barriers compromised by topical tacrolimus. J Invest Dermatol. 2011 Mar;131(3):698-705. doi: 10.1038/jid.2010.344. Epub 2010 Nov 25. PMID 21107352
- [Background] Jiang YJ, Lu B, Crumrine D, Elias PM, Feingold KR. IL-6 stimulates but is not essential for stratum corneum formation and permeability barrier development during gestation. Exp Dermatol. 2010 Aug;19(8):e31-6. doi: 10.1111/j.1600-0625.2009.00968.x. PMID 19758319
- [Background] Upragarin N, Landman WJ, Gaastra W, Gruys E. Extrahepatic production of acute phase serum amyloid A. Histol Histopathol. 2005 Oct;20(4):1295-307. doi: 10.14670/HH-20.1295. PMID 16136510
- [Background] Constantin MM, Poenaru E, Poenaru C, Constantin T. Skin Hydration Assessment through Modern Non-Invasive Bioengineering Technologies. Maedica (Bucur). 2014 Mar;9(1):33-8. PMID 25553123
- [Background] Mundelein M, Valentin B, Chabicovsky R, et al. Transepidermal water loss (TEWL) measurements with two novel sensors based on different sensing principles. Sensors and Actuators A Physical 2007;142(1): DOI 10.1016/j.sna.2007.04.012
- [Background] Pinnagoda J, Tupker RA, Agner T, Serup J. Guidelines for transepidermal water loss (TEWL) measurement. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1990 Mar;22(3):164-78. doi: 10.1111/j.1600-0536.1990.tb01553.x. PMID 2335090
- [Background] Kottner J, Lichterfeld A, Blume-Peytavi U. Transepidermal water loss in young and aged healthy humans: a systematic review and meta-analysis. Arch Dermatol Res. 2013 May;305(4):315-23. doi: 10.1007/s00403-012-1313-6. Epub 2013 Jan 23. PMID 23341028